CLINICAL TRIAL: NCT01772719
Title: Overcoming Chemotherapy Resistance In Refractory Multiple Myeloma With Simvastatin and Zoledronic Acid
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left institution-study not continued
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCC-HEM-11-003
Record Dates: First submitted 2011-11-15; First posted 2013-01-21 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Multiple Myeloma
Keywords: refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Simvastatin; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Arm (Experimental): Study Arm
  Interventions: Drug: Simvastatin and zoledronic acid

INTERVENTIONS:
Drug: Simvastatin and zoledronic acid — 1. Simvastatin 80 mg PO daily starting two days before starting chemotherapy and stopping two days after chemotherapy.
  2. Zoledronic acid 4 mg IV over 15 minutes on day 1 and then monthly.
  Other Names: Zocor

SUMMARY:
The purpose of this study is to examine the effect of simvastatin and zoledronic acid on M-protein and/or free light chains when added to conventional chemotherapy for the treatment of multiple myeloma patients.

DETAILED DESCRIPTION:
We hypothesize that the addition of simvastatin and zoledronic acid to bortezomib, thalidomide, melphalan or dexamethasone based regimens will decrease drug resistance when treating refractory multiple myeloma. We hypothesize that the addition of simvastatin and zoledronic acid will not increase the chemotherapy toxicity significantly and will be tolerable for patients. We believe simvastatin and zoledronic acid have antitumor properties and will contribute to reversal of resistance. Treatment will be significantly enhanced when these agents are combined

ELIGIBILITY:
Inclusion Criteria:

1. have a definitive diagnosis of Multiple Myeloma (using the International Myeloma Working Group Guidelines).
2. meet one of the following two requirements:

   * Have achieved minimal response (MR) or stable disease (SD) in current treatment regimen after a minimum of two cycles.
   * Have partial response but show no further improvement in paraprotein levels in the latest two measurements.
3. must have measurable active or symptomatic disease. Measurable disease may be paraprotein or free light chains in serum or urine, or the presence of bone marrow plasma cells, defined by one or more of the following criteria:

   * Presence of serum M-protein concentration > 1g/dL.
   * Urine M-protein excretion > 200mg in 24-hour urine collection.
   * Serum free light chain concentration ≥ 10mg/dL and abnormal kappa/lambda ratio.
   * Urine free light chain concentration ≥ 100mg/L and abnormal kappa/lambda ratio.
   * Bone marrow plasma cell percentage ≥ 30% (if no detectable M-protein or FLC.)
4. Age > 18 years of age.
5. If female with reproductive capacity: on effective means of birth control during the entire duration of the treatment.
6. Patients must have recovered from acute toxicities resulting from therapy administered prior to entering this study to grade 1 or less (CTCAE 4) Alopecia may not be resolved.
7. Ability to understand and willingness to sign a written informed consent document.
8. Life expectancy of greater than 8 weeks.
9. ECOG performance status 0, 1, or 2 (Karnofsky > 60%; see Appendix A).
10. have adequate bone marrow function as defined below:

    * absolute neutrophil count > 500/ul
    * platelets > 30,000/ul
11. have adequate liver function as defined below:

    * total bilirubin < 2 times the upper limit of normal
    * AST(SGOT), ALT(SGPT) < 3 x upper limit of normal
12. have adequate renal function as defined by a creatinine clearance > 40 mL/min (measured or estimated by the Cockcroft-Gault formula).
13. have no signs of significant rhabdomyolysis determined by CPK levels with a CK < 5 times the upper limit of normal.

Exclusion Criteria:

1. have not received any chemotherapy treatment for multiple myeloma prior to being enrolled in the study.
2. show progressive disease or are not tolerating current chemotherapy regimen.
3. were receiving simvastatin (dose > 40mg/day) while receiving current chemotherapy regimen for multiple myeloma.
4. failed or progressed on more than two chemotherapy regimens, including current treatment; prior to enrolling in this study.
5. receiving any other investigational agent(s).
6. Active second malignancy in the last 5 years except for non-melanoma skin cancer or carcinoma-in-situ.
7. Pregnant women are ineligible, as treatment involves unforeseeable risks to the embryo or fetus. Female patients with reproductive capacity are required to use effective means of birth control during the entire duration of the treatment.
8. History of hypersensitivity reactions attributed to simvastatin or zoledronic acid.
9. receiving medications that may increase risk of rhabdomyolysis such as itraconazole, ketoconazole, erythromycin, cyclosporine, amiodarone, verapamil, clarithromycin, nefazodone, ranolazine, HIV protease inhibitors, gemfibrozil, posaconazole, danazol, amiodarone, diltiazem and amlodipine.
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, myopathy, untreated hypothyroidism, hereditary myopathy in the family history, unstable angina pectoris, liver disease not due to multiple myeloma, cardiac arrhythmia that is symptomatic or not rate controlled, active connective tissue disease, active autoimmune disease, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Rodriguez, MD, Principal Investigator — Dept. of Med Admin.
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 7 subjects were enrolled into this trial by the investigator from medical clinic
Period: Overall Study
Arm/Group | Simvastatin and Zoledronic Acid
Started | 7
Completed | 0
Not Completed | 7
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Study Arm: Study Arm
  Simvastatin and zoledronic acid: 1. Simvastatin 80 mg PO daily starting two days before starting chemotherapy and stopping two days after chemotherapy.
  2. Zoledronic acid 4 mg IV over 15 minutes on day 1 and then monthly.
Arm/Group | Study Arm
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 63 [53 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Paraprotein Level and Free Light Chain (FLC) Ratio From Baseline Measurement
Description: The effect of simvastatin and zolendronic acid on M-Protein and FLC ratio will be measured 4 weeks after treatment begins, then every 4 weeks until progression of disease.
Time Frame: 4 weeks after treatment begins
Population: NA = Not available, Study was terminated and PI has left the institution. Sincere efforts were made to gather and report the data, however, no data is available for the study
Groups:
- Simvastatin and Zolendronic Acid: Simvastatin and zoledronic acid:
  1. Simvastatin 80 mg PO daily starting two days before starting chemotherapy and stopping two days after chemotherapy.
  2. Zoledronic acid 4 mg IV over 15 minutes on day 1 and then monthly.
Arm/Group | Simvastatin and Zolendronic Acid
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Survival
Description: OS(Overall survival) is measured from date of study enrollment until death.
Time Frame: At start of year 2 of follow-up on all surviving participants
Population: Study was terminated and PI has left the institution. Sincere efforts were made to gather and report the data, however, no data is available for the study
Arm/Group | Simvastatin and Zoledronic Acid
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response
Description: Response will be accessed by one of the study investigators at each monthly follow up visit during year one.
Time Frame: Year 1 follow up visits occur monthly
Population: Study Terminated, zero total participants analyzed
Arm/Group | Simvastatin and Zoledronic Acid
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Study will estimate PFS when there is one year of follow up data for all surviving participants
Time Frame: At start of year 2 follow up on all surviving participants
Population: as for outcome 2
Arm/Group | Simvastatin and Zoledronic Acid
Number analyzed (Participants) | 0

5. Secondary Outcome: Duration of Response
Description: Response will be assessed by one of the study investigators at each three month follow up visit for Year 2
Time Frame: Year 2 follow up visit occur every three months
Population: as for outcome 2
Arm/Group | Simvastatin and Zoledronic Acid
Number analyzed (Participants) | 0

6. Secondary Outcome: Duration of Response
Description: Response will be assessed by one of the study investigators at each six month follow up visit for Year 3-5
Time Frame: Year 3-5 follow up visit occurs every six months
Population: as for outcome 2
Arm/Group | Study Arm
Number analyzed (Participants) | 0

7. Secondary Outcome: Incidence Rate of Toxicity
Description: Descriptive statistics will be provided regarding incidence rates of toxicity. Patients will be monitored for safety throughout the study.
Time Frame: Every 12 months up to one month after treatment completion
Population: as for outcome 2
Arm/Group | Simvastatin and Zoledronic Acid
Number analyzed (Participants) | 0

8. Secondary Outcome: Comparison of Quality of Life Scores
Description: The QOL scores taken at the start of the study and every 4 months after treatment starts will be analyzed using Wilcoxon test for paired differences
Time Frame: Up to 2 months after last treatment has been completed
Population: as for outcome 2
Arm/Group | Simvastatin and Zoledronic Acid
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Study Arm
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes